CLINICAL TRIAL: NCT01853579
Title: Thyroid Hormone Replacement for Subclinical Hypothyroidism (TRUST) - Subanalysis on Subclinical Hypothyroidism and Depression
Brief Title: The TRUST Study - Depression Substudy
Acronym: TRUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Leiden University Medical Center (Other); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 162/11; 2011-004554-26 (Registry Identifier: EudraCT); 01660126 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2013-05-06; First posted 2013-05-15 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Subclinical Hypothyroidism; Depression
Keywords: Randomized controlled trial; Subclinical hypothyroidism; Levothyroxine; Depression
MeSH Terms: conditions — Depression | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Experimental: Drug: Levothyroxine The intervention will start with Levothyroxine 50 mcg daily (reduced to 25 mcg in subjects <50 kg of body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) vs. matching placebo; at 3 months, if the serum TSH level is <0.4 mU/L, dose will be reduced by 25 mcg; TSH >=0.4 and <4.6 mU/L, no change to dose; TSH >=4.6 mU/L, additional 25 mcg. The process will be repeated at 12 months, then annually; mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine which will be prescribed is 150 mcg (after 4 increments of 25 mcg at 3 months, 1, 2, 3 years; from the starting dose of 50 mcg).
  Interventions: Drug: Levothyroxine
- 2 (Placebo Comparator): Placebo Comparator: Drug: Placebo Control patients will obtain a placebo pill of the same characteristics as the intervention drug, and mock titration will be carried out identically to the intervention drug.
  Pharmaceutical composition of placebo (100 mg): Lactose monohydrate 66 mg, Maize starch 25 mg, Gelatin 5 mg, Croscarmellose sodium 3.5 mg, Magnesium stearate (vegetable source) 0.5 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxine — The intervention will start with Levothyroxine 50 µg daily (reduced to 25 µg in subjects <50Kg body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) versus matching placebo; at 3 months if the serum TSH level is <0.4 mU/L dose will be reduced by 25 µg; TSH >=0.4 and <4.6 mU/L, no change to dose; TSH >=4.6mUL, additional 25 µg. The process will be repeated at 12 months then annually. Mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine that will be prescribed is 150μg (after 4 increments of 25μg at 3 months, 1, 2 and 3 years; from the starting dose of 50μg).
  Arms: 1
Drug: Placebo — Control patients will obtain a placebo pill of the same characteristics as the intervention drug, and mock titration will be carried out identically to the intervention drug.
  Pharmaceutical composition of placebo (100 mg): Lactose monohydrate 66 mg, Maize starch 25 mg, Gelatin 5 mg, Croscarmellose sodium 3.5 mg, Magnesium stearate (vegetable source) 0.5 mg.
  Arms: 2

SUMMARY:
Mild thyroid failure is a common condition among older adults and has been associated with numerous adverse effects on health, such as cardiovascular disease, cognition disturbances and muscular problems. Mild thyroid failure has also been associated with an increased risk of developing depression. To date, only few studies have investigated the effect of thyroid hormone replacement on depression in patients with mild thyroid failure. This study therefore aims to assess whether thyroid hormone replacement in older adults with mild thyroid failure is associated with a decrease in the presence of depressive symptoms. This study forms a substudy of a large international study on thyroid hormone replacement in older adults with mild thyroid failure (the TRUST study).

DETAILED DESCRIPTION:
Background

Subclinical hypothyroidism is a common condition among older adults, particularly above the age of 65 years, with a prevalence reaching 10 to 15% of the population. This condition has been associated with numerous adverse outcomes, such as cardiovascular disease, cognition disturbances and muscular problems. All of these potential outcomes will be assessed in the TRUST study. Subclinical hypothyroidism has also been associated with an increased risk of developing depression. It has been suggested that subclinical hypothyroidism may lower the threshold for the development of depression. The prevalence of depression among community-dwelling elderly ranges from 2 to 10%. Patients with depression have been shown to have a lower response to anti-depressive drugs when they have subclinical hypothyroidism. Only a few randomized studies in patients with subclinical hypothyroidism have studied the effect of thyroid hormone replacement on depression, with conflicting results: the studied populations were often small (maximal number of participants: 143), using different scales to measure the presence of depressive symptoms.

Objective

To investigate whether thyroid hormone replacement in older adults with subclinical hypothyroidism is associated with a decrease in the presence of depressive symptoms in a sub-study of the TRUST study.

Methods Use of the 15-item Geriatric Depression Scale (GDS-15) to measure depressive symptoms in all 450 patients included in the TRUST study in Switzerland and the Netherlands, the most validated test for depression screening, with validity to measure longitudinal changes. GDS-15 will be applied at baseline and after 1 year to compare changes in depression scores between placebo and thyroxin arms. Power calculation (ANCOVA method) with 225 participants per treatment group, assuming a standard deviation of 3 and a baseline to follow up correlation of 0.7, results in 99.9% power for detecting a mean difference of 1.0 points at a two-sided alpha-level of 0.05. Depending on recruitment for the main trial (ClinicalTrials.gov ID: NCT01660126) in respective countries, a lower number of participants may be included, retaining a very large power for this continuous outcome.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling patients aged >= 65 years with subclinical hypothyroidism
* Written informed consent

Exclusion Criteria

* Subjects currently on Levothyroxine or antithyroid drugs, amiodarone or lithium
* Recent thyroid surgery or radio-iodine (within 12 months)
* Grade IV NYHA heart failure
* Prior clinical diagnosis of dementia
* Recent hospitalisation for major illness or elective surgery (within 4 weeks)
* Terminal illness
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects who are participating in ongoing RCTs of therapeutic interventions (including CTIMPs)
* Plan to move out of the region in which the trial is being conducted within the next 2 years (proposed minimum follow-up period)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 426 (Actual)
Dates: Start 2013-03; Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 15-items Geriatric Depression Scale | At 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, MD, MAS, Principal Investigator — University Clinic of General Internal Medicine, Bern University Hospital, Bern, Switzerland; Jacobijn Gussekloo, MD, Principal Investigator — Leiden University Medical Center, Leiden, The Netherlands
Locations (3):
- Leiden University Medical Center, Leiden, Netherlands
- Switzerland (2):
  - Department of General Internal Medicine, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern

REFERENCES:
- [Derived] Wildisen L, Feller M, Del Giovane C, Moutzouri E, Du Puy RS, Mooijaart SP, Collet TH, Poortvliet RKE, Kearney P, Quinn TJ, Kloppel S, Bauer DC, Peeters RP, Westendorp R, Aujesky D, Gussekloo J, Rodondi N. Effect of Levothyroxine Therapy on the Development of Depressive Symptoms in Older Adults With Subclinical Hypothyroidism: An Ancillary Study of a Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e2036645. doi: 10.1001/jamanetworkopen.2020.36645. PMID 33566107